CLINICAL TRIAL: NCT05676424
Title: Assessment of the Cognitive Load of the Landed Combatant in Virtual Reality.
Acronym: ECCOREV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PBMD07; 2022-A01311-42 (Other: IDRCB)
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Fatigue
Keywords: cognitive overload
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To support the landed soldier during operational missions in hostile environment, equipment must be designed to enable soldiers to cope with strong visual, auditory and informational demands. Technological solutions proposed by manufacturers are embodied in increasingly sophisticated systems.

These systems take too little account of the characteristics of the perceptive and cognitive skills of human beings in an action situation.

Cognitive load results from the interaction between, on the one hand, the characteristics of the task and the constraints it imposes, and on the other hand, the resources available to the individual, in terms of skills, motivation, physiological state and social support. The phenomenon of cognitive overload occurs when the individual no longer has sufficient resources to meet the demands of the task, which leads to a deterioration in his performance which, in high-risk situations, jeopardizes his safety.

Tasks are treated differently depending on their level of difficulty. We will base ourselves on Rasmussen's SRK (Skill Rule Knowledge) model, which describes three levels of information processing: level S refers to the (automatic) processing of sensory-motor and cognitive skills, level R refers to the execution of rules and procedures embedded in mental models, and level K refers to the mental activities of elaborating procedures, based on high-level cognitive mechanisms, such as anticipation, evaluation or planning. Multitasking situations are therefore generally composed of tasks of various levels of difficulty which lead to a higher or lower cost of cognitive control.

Thus, this study is aimed at identifying variations in the subjective level of cognitive load of landed combatants (group leaders) as a function of the level of difficulty of primary tasks.

ELIGIBILITY:
Inclusion Criteria:

* to be a soldier in an infantry regiment,
* to be a group leader.

Exclusion Criteria:

* to be in a situation of motor disability,
* to have a cardiac pathology,
* to have a visual pathology not corrected by glasses or contact lenses,
* to have a hearing impairment,
* to have a psychiatric disorder; a progressive neurological or organic pathology requiring drug treatment,
* to take psychotropic drugs,
* to take more than 28 units of alcohol per week,
* to be epileptic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is composed of healthy soldiers serving as group leaders in an infantry regiment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Subjective level of cognitive load, measured with the National Aeronautics and Space AdministrationTask Load Index (NASA-TLX) | Through study completion (12 months)
  The National Aeronautics and Space AdministrationTask Load Index (NASA-TLX) is a widely used, subjective, multidimensional assessment tool that rates perceived workload in order to assess a task, system, or team's effectiveness or other aspects of performance.
  The NASA-TLX score is comprised between 0 and 100 with higher score meaning high level of cognitive load.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided